CLINICAL TRIAL: NCT04162873
Title: RESILIENCE: Effect of Comprehensive Celecoxib Through Treatment for Advanced-Stage Head and Neck Cancer: A Randomized, Double-Blinded, Placebo-Controlled Trial
Brief Title: Celecoxib Through Surgery and Radiation Therapy for the Treatment of Advanced Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HCI124211; NCI-2019-07104 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HCI124211 (Other: Huntsman Cancer Institute/University of Utah); P30CA042014 (NIH)
Record Dates: First submitted 2019-11-04; First posted 2019-11-14 (Actual); Results first posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Clinical Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage IV HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Nasal Cavity and Paranasal Sinus Carcinoma; Oral Cavity Carcinoma; Pathologic Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Pathologic Stage IV HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Recurrent Hypopharyngeal Carcinoma; Recurrent Laryngeal Carcinoma; Recurrent Nasal Cavity and Paranasal Sinus Carcinoma; Recurrent Oral Cavity Carcinoma; Recurrent Oropharyngeal Carcinoma; Stage III Hypopharyngeal Carcinoma AJCC v8; Stage III Laryngeal Cancer AJCC v8; Stage III Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IV Hypopharyngeal Carcinoma AJCC v8; Stage IV Laryngeal Cancer AJCC v8; Stage IV Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IVA Hypopharyngeal Carcinoma AJCC v8; Stage IVA Laryngeal Cancer AJCC v8; Stage IVA Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IVB Hypopharyngeal Carcinoma AJCC v8; Stage IVB Laryngeal Cancer AJCC v8; Stage IVB Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IVC Hypopharyngeal Carcinoma AJCC v8; Stage IVC Laryngeal Cancer AJCC v8; Stage IVC Oropharyngeal (p16-Negative) Carcinoma AJCC v8
MeSH Terms: conditions — Oropharyngeal Neoplasms; Paranasal Sinus Neoplasms; Mouth Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Carcinoma | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Celecoxib Arm (Experimental): Patients receive celecoxib PO or via feeding tube BID starting 1 to 7 days prior to surgery and continues until the completion of radiation therapy (up to 6 months in total) in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Celecoxib; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Placebo Arm (Placebo Comparator): Patients receive placebo PO or via feeding tube BID starting 1 to 7 days prior to surgery and continues until the completion of radiation therapy (up to 6 months in total) in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Placebo; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Celecoxib — Given PO or via feeding tube
  Other Names: Benzenesulfonamide, 4-[5-(4-methylphenyl)-3-(trifluoromethyl)-1H-pyrazol-1-yl]-; Celebrex; SC-58635; YM 177
  Arms: Celecoxib Arm
Other: Placebo — Given PO or via feeding tube
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Placebo Arm
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well celecoxib works through surgery and radiation therapy in treating patients with head and neck cancer that has spread to other places in the body (advanced). Celecoxib is Food and Drug Administration approved to treat arthritis, acute pain, and painful menstrual periods. Adding celecoxib to standard of care treatment may help to decrease the amount of time between surgery and radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the number of days from surgery to initiation of radiation with the addition of celecoxib compared to placebo.

SECONDARY OBJECTIVES:

I. To assess overall pain control and management for patients on celecoxib compared to placebo.

* Subjective pain scores on the visual analog scale of pain intensity averaged over a week at rest, with a swallow, and with a cough.
* Patient satisfaction with pain control questionnaire.
* Narcotic consumption in daily total morphine equivalents averaged over a week. II. To assess functional outcomes for patients on celecoxib compared to placebo.

III. To assess the effect of celecoxib therapy on Quality of Life (QoL) compared to placebo.

IV. To assess the average number of treatment days missed during adjuvant radiation for patients on celecoxib compared to placebo.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive celecoxib orally (PO) or via feeding tube twice daily (BID) starting 5 days prior to surgery and continues until the completion of radiation therapy (up to 6 months in total) in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive placebo PO or via feeding tube BID starting 5 days prior to surgery and continues until the completion of radiation therapy (up to 6 months in total) in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged ≥ 18 years.
* Advanced-stage (overall stage III and IV) head and neck cancers (sinonasal oral cavity, oropharynx, larynx, and hypopharynx) undergoing surgical resection and then adjuvant radiation. Primary and recurrence cases are acceptable
* Karnofsky performance status of >= 70
* Hemoglobin >= 10 g/dL
* Total bilirubin =< 2 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal (ULN)
* Albumin > 3.5 g/dL
* Estimated glomerular filtration rate (eGFR) >= 30 mL/min/1.73 m^2 or creatinine clearance >= 30 mL/min by Cockcroft-Gault
* Serum potassium within normal limits
* Negative serum or urine pregnancy test at screening for women of childbearing potential
* Highly effective contraception for female subjects throughout the study and for at least 5 days after the last dose of study therapy if the risk of conception exists
* Recovery to baseline or =< grade 1 Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy
* Willing to maintain a diary of all opioids used during the trial for the treatment of pain
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines
* Subject has verbally confirmed they are willing to complete adjuvant radiation therapy if recommended after surgery per protocol.
* Adjuvant radiation has been recommended by the institutional treatment planning conference with the best available data, but will be confirmed based on final surgical pathology.

Exclusion Criteria:

* Known distant metastatic disease or the tumor is deemed not surgically resectable
* Established in a pain management clinic or has taken opioids regularly >= 6 months
* Known or suspected to be poor CYP2C9 metabolizers based on previous history/experience with other CYP2C9 substrates (such as warfarin, phenytoin)
* Known hypersensitivity to celecoxib, aspirin, other non-steroidal anti-inflammatory drug (NSAID)s, or sulfonamides
* Uncontrolled hypertension defined as blood pressure (BP) > 150 mmHg systolic or > 90 mmHg diastolic on three consecutive reads, taken in one sitting despite optimal antihypertensive treatment
* Patients with a known history of the following:

  * Cerebrovascular accident (CVA), stroke, or cardiovascular thrombotic events (e.g. acute myocardial infarction).
  * Chronic heart failure.
  * Gastrointestinal bleeding, ulceration, peptic ulcer disease, or perforation of the stomach or intestines.
  * Aspirin-sensitive asthma.
  * Chronic kidney disease, stage 4 or 5
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* The subject has uncontrolled, significant intercurrent or recent illness requiring systemic therapy, would preclude safe study participation, or is deemed clinically significant by the investigator
* Known human immunodeficiency virus (HIV) infection with a detectable viral load within 6 months of the anticipated start of treatment.

  * Note: Patients on effective anti-retroviral therapy with an undetectable viral load within 6 months of the anticipated start of treatment are eligible for this trial
* Known chronic hepatitis B virus (HBV) or hepatitis C virus infection with a detectable viral load.

  * Note: Patients with an undetectable HBV viral load on appropriate suppressive therapy are eligible. Patients with an undetectable hepatitis C virus (HCV) viral load on appropriate treatment are eligible
* Subjects taking prohibited medications . A washout period of prohibited medications for a period of at least 5 half-lives or as clinically indicated should occur prior to the start of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Cannon, MD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 13 participants were enrolled in the study. One participant withdrew from the study prior to receiving the first dose of study drug.
Groups:
- Celecoxib Arm: Patients received celecoxib PO or via feeding tube BID starting 1 to 7 days prior to surgery and continued until the completion of radiation therapy (up to 6 months in total) in the absence of disease progression or unacceptable toxicity.
  Celecoxib: Given PO or via feeding tube
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
- Placebo Arm: Patients received placebo PO or via feeding tube BID starting 1 to 7 days prior to surgery and continued until the completion of radiation therapy (up to 6 months in total) in the absence of disease progression or unacceptable toxicity.
  Placebo: Given PO or via feeding tube
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
Period: Overall Study
Arm/Group | Celecoxib Arm | Placebo Arm
Started | 5 | 7
Completed | 4 | 7
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Celecoxib Arm | Placebo Arm | Total
Number analyzed (Participants) | 5 | 7 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 2 | 5 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.40 (7.02) | 65.14 (20.24) | 63.17 (15.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 2 | 6 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 4 | 6 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 7 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 7 | 12
Initial Histologic Grade [Count of Participants; unit: Participants] — Staging systems are utilized in cancer care to standardize the extent of cancer. The TNM (Tumor, Nodes, Metastasized) system is used for squamous cell carcinomas.
  With this system, G describes the grade of the cancer. The grade score is based on Differentiation (1-Normal cells to 3-Very abnormal cells), Mitotic count (1 to 3; low score means fewer cells were dividing), and Tumor necrosis (0 to 2; lower score means less dying tissue).
  This has possible scores of GX (grade cannot be assessed due to incomplete information), G1 (score of 2-3), G2 (score of 4-5), and G3 (score of 6-8).
  Participants
    Gx | 0 | 0 | 0
    G1 | 3 | 3 | 6
    G2 | 2 | 4 | 6
    G3 | 0 | 0 | 0
Prognostic Stage [Count of Participants; unit: Participants] — Staging systems are utilized to standardize the extent of cancer, and the TNM (Tumor, Nodes, Metastasized) system is used for squamous cell carcinomas.
  The TNM status is tabulated to give a numerical status from Stage I (T1, N0, and M0) to Stage IVC (any T, any N, and M1).
  Participants
    Stage III | 2 | 2 | 4
    Stage IVA | 3 | 5 | 8
    Stage IVB | 0 | 0 | 0
    Stage IVC | 0 | 0 | 0
Type of Head and Neck Cancer [Count of Participants; unit: Participants]
  Hypopharynx | 0 | 0 | 0
  Larynx | 0 | 0 | 0
  Oral Cavity | 5 | 6 | 11
  Oropharynx | 0 | 0 | 0
  Sinonasal | 0 | 1 | 1
Primary or Recurrent Tumor [Count of Participants; unit: Participants]
  Primary | 4 | 7 | 11
  Recurrent | 1 | 0 | 1
Laterality [Count of Participants; unit: Participants]
  Right | 2 | 0 | 2
  Left | 2 | 6 | 8
  Center/Both | 1 | 1 | 2
Primary Tumor pT [Count of Participants; unit: Participants] — Staging systems are utilized in cancer care to standardize the extent of the cancer. The TNM (Tumor, Nodes, Metastasized) system is used for bladder cancer.
  With this system, T describes how far the primary tumor has grown and if it has grown into nearby tissue. This staging system ranges from T0 (No evidence of a primary tumor), T4a (tumor has grown beyond a certain point; moderately advanced), to T4b (tumor has grown further than T4a; very advanced).
  Participants
    pT1 | 1 | 0 | 1
    pT3 | 1 | 1 | 2
    pT4a | 3 | 4 | 7
    rpT4a | 0 | 1 | 1
    mpT3 | 0 | 1 | 1
Regional Lymph Nodes pN [Count of Participants; unit: Participants] — Staging systems are utilized in cancer care to standardize the extent of the cancer. The TNM (Tumor, Nodes, Metastasized) system is used for squamous cell carcinomas. With this system, N describes if any cancer spread to lymph nodes.
  This staging system ranges from NX (cannot be assessed), N0 (no regional lymph node spread), N2a (cancer has spread to a single lymph node on the same side of the body as the primary tumor), N2b (cancer has spread to multiple lymph nodes on the same side of the body), to N3b (tumor extends to the supraclavicular fossa).
  Participants
    pN0 | 0 | 4 | 4
    pN2a | 1 | 0 | 1
    pN2b | 1 | 0 | 1
    pN3b | 2 | 1 | 3
    pNx | 1 | 0 | 1
    N2b | 0 | 1 | 1
    rpN0 | 0 | 1 | 1
Distant Metastasis pM [Count of Participants; unit: Participants] — Staging systems are utilized in cancer care to standardize the extent of the cancer. The TNM (Tumor, Nodes, Metastasized) system is used for squamous cell carcinomas. With this system, M describes if any cancer spread to other parts of the body.
  This staging system ranges from MX (Cancer spread cannot be assessed), M0 (cancer has not spread), to M1 (cancer has spread).
  Participants
    pM0 | 1 | 1 | 2
    pMx | 3 | 3 | 6
    rpMx | 0 | 1 | 1
    Mx | 0 | 1 | 1
    Not Applicable | 1 | 1 | 2
KPS Score [Count of Participants; unit: Participants] — Assessment of current activity level was assessed utilizing Karnofsky Performance Status (KPS). The KPS is a scale used to measure a subject's ability to perform daily tasks from 100 Normal no complaints no evidence of disease, 50 Requires considerable assistance and frequent medical care, and 0 Dead.
  Participants
    100 - Normal; no complaints; no evidence of disease | 1 | 0 | 1
    90 - Able to carry on normal activity; minor signs or symptoms of disease | 3 | 6 | 9
    80 - Normal activity with effort; some signs or symptoms of disease | 1 | 1 | 2
Functional Oral Intake Scale [Count of Participants; unit: Participants] — Assessment of current activity level was assessed utilizing Functional Oral Intake Scale (FOIS).
  FOIS is a standardized scale assessed by the treating investigator to determine the functional level of oral intake in patients with dysphagia. The FOIS measures from 1 (Aspirates saliva, Nothing by mouth), 2 (Tube dependent, Nothing by mouth/minimal trials), 3 (Tube dependent, Full trials by mouth), 4 (Total Oral Single, texture trials), 5 (Total Oral, Multiple texture trials), 6 (Total Oral, By mouth/ restrictions Minimal), and 7 (Regular diet, By mouth/ no restrictions).
  Participants
    3 - Tube Dependent (full trials by mouth) - Severe Deficit | 0 | 1 | 1
    5 - Total Oral (multiple texture trials) - Mild Deficit | 3 | 0 | 3
    6 - Total Oral (by mouth/restrictions) - Minimal Deficit | 2 | 5 | 7
    7 - Regular Diet (by mouth/no restrictions) - Normal | 0 | 1 | 1
Feeding Tube [Count of Participants; unit: Participants]
  Yes | 0 | 1 | 1
  No | 5 | 6 | 11
Height [Mean (Standard Deviation); unit: cm] | 170.68 (8.55) | 177.66 (11.34) | 174.75 (10.47)
Weight [Mean (Standard Deviation); unit: kg] | 83.12 (20.44) | 85.63 (21.10) | 84.58 (19.91)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.20 (4.95) | 26.95 (4.83) | 27.47 (4.69)
Pulse [Mean (Standard Deviation); unit: bpm] | 76.40 (7.70) | 84.14 (21.43) | 80.92 (16.97)
Blood Pressure [Mean (Standard Deviation); unit: mmHg]
  Systolic | 118.20 (11.92) | 135.71 (12.39) | 128.42 (14.72)
  Diastolic | 77.20 (6.72) | 77.71 (7.63) | 77.50 (6.95)
Respiratory Rate [Mean (Standard Deviation); unit: Breaths per Minute] | 18 (1.41) | 16 (1.15) | 16.83 (1.59)
Temperature [Mean (Standard Deviation); unit: Fahrenheit] | 97.98 (0.51) | 97.98 (0.52) | 97.98 (0.49)
Assessment of Overall Pain Control and Management for Patients [Count of Participants; unit: Participants] — Patient satisfaction was assessed with a pain control questionnaire. The participants were asked how satisfied they were with their overall pain control over the last seven days. Satisfaction was measured from (0) Very Dissatisfied to (4) Very satisfied.
  Participants
    Not Assessed | 0 | 1 | 1
    0) Very Dissatisfied | 0 | 1 | 1
    1) Somewhat dissatisfied | 3 | 0 | 3
    2) Neutral | 1 | 1 | 2
    3) Somewhat satisfied | 1 | 1 | 2
    4) Very satisfied | 0 | 3 | 3
Visual Analog Scale [Count of Participants; unit: Participants] — Assessment of subjective pain scores on the visual analog scale of pain intensity averaged over a week at rest, with a swallow, and with a cough. The subjects rated their pain from 0-10 on the pain intensity scale. Scores are reported as No Pain (0), Mild Pain (0.5-4.4), Moderate Pain (4.5-7.4), and Severe Pain (7.5-10).
  Participants
    While at Rest: No Pain (0-0.5) | 1 | 3 | 4
    While at Rest: Mild Pain (0.5-4.4) | 1 | 2 | 3
    While at Rest: Moderate Pain (4.5-7.4) | 3 | 2 | 5
    While at Rest: Severe Pain (7.5-10) | 0 | 0 | 0
    With a Swallow: No Pain (0-0.5) | 1 | 2 | 3
    With a Swallow: Mild Pain (0.5-4.4) | 2 | 3 | 5
    With a Swallow: Moderate Pain (4.5-7.4) | 1 | 1 | 2
    With a Swallow: Severe Pain (7.5-10) | 1 | 1 | 2
    With a Cough: No Pain (0-0.5) | 1 | 3 | 4
    With a Cough: Mild Pain (0.5-4.4) | 2 | 4 | 6
    With a Cough: Moderate Pain (4.5-7.4) | 1 | 0 | 1
    With a Cough: Severe Pain (7.5-10) | 1 | 0 | 1
European Organization for Research &Treatment of Cancer Quality of Life Head & Neck (EORTC QLQ-HN43) [Mean (Standard Deviation); unit: units on a scale] — EORTC QLQ-HN43 is a 43-question survey of health-related quality of life of cancer patients assessing symptoms in the past week from "1 Not at All" to "4 Very Much".
  Scores are from 0-100; high scores represent a high response. A high functional scale score (FS; body image, social contact, &sexuality) represent a high level of function.
  A high symptom scale score (SS; anxiety, cough, pain, swallow, neurologic problems, senses, speech, social eating, weight loss, problems w/ skin, shoulder, wound healing, dry mouth, opening mouth, neck swelling, &teeth) represent a high level of symptoms
  units on a scale
    Anxiety (SS) | 70.0 (24.72) | 59.52 (33.13) | 63.89 (29.16)
    Body Image (FS) | 46.67 (36.35) | 92.06 (8.40) | 73.15 (32.64)
    Coughing (SS) | 26.67 (27.89) | 4.76 (12.60) | 13.89 (22.29)
    Dry mouth and sticky saliva (SS) | 36.67 (27.39) | 21.43 (15.85) | 27.78 (21.71)
    Neurological Problems (SS) | 13.33 (29.81) | 4.76 (12.60) | 8.33 (20.72)
    Opening mouth (SS) | 66.67 (33.33) | 28.57 (29.99) | 44.44 (35.77)
    Pain in the head and neck (SS) | 66.67 (27.64) | 38.10 (26.29) | 50.00 (29.52)
    Social Contact (FS) | 46.67 (44.72) | 95.24 (12.60) | 75.00 (37.94)
    Problems with senses (SS) | 20 (27.39) | 4.76 (8.13) | 11.11 (19.25)
    Skin Problems (SS) | 15.56 (21.66) | 3.17 (8.40) | 8.33 (15.80)
    Swelling in the neck (SS) | 53.33 (38.01) | 19.05 (26.23) | 33.33 (34.82)
    Social Eating (SS) | 63.33 (27.39) | 22.62 (20.25) | 39.58 (30.59)
    Speech Problems (SS) | 62.67 (36.70) | 24.76 (35.43) | 40.56 (39.44)
    Problems with Swallowing (SS) | 48.33 (35.06) | 15.48 (18.90) | 29.17 (30.46)
    Problems with Sexuality (FS) | 50.00 (47.14) | 66.67 (42.16) | 59.09 (43.05)
    Problems with teeth (SS) | 51.11 (30.02) | 22.22 (19.25) | 34.26 (27.40)
    Weight loss (SS) | 26.67 (43.46) | 23.81 (31.71) | 25 (35.18)
    Problems with Wound Healing (SS) | 20 (29.81) | 28.57 (40.50) | 25.00 (35.18)
    Shoulder Problems (SS) | 13.33 (29.81) | 0 (0) | 5.56 (19.25)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Days From Surgery to the Initiation of Radiation and Adjuvant Therapy
Description: The day of surgery will be considered day 0 and the number of days will be counted until the first dose of adjuvant radiation. This outcome measure will report the mean number of days from surgery to the initiation of radiation and adjuvant therapy for the Celecoxib and Placebo Arms.
Time Frame: up to 3 months
Population: Two participants in the Celecoxib Arm did not receive adjuvant radiation therapy and were not evaluable for this endpoint. One other participant from the Celecoxib Arm only received two doses of study treatment and was not evaluable for this endpoint.
  One participant in the Placebo Arm did not receive adjuvant radiation therapy and was not evaluable for this endpoint.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Celecoxib Arm | Placebo Arm
Number analyzed (Participants) | 2 | 6
days | 53.5 (9.19) | 60.17 (20.04)

2. Secondary Outcome: Assessment of Overall Pain Control and Management for Patients on Celecoxib Compared to Placebo - Visual Analog Scale.
Description: Assessment of subjective pain scores on the visual analog scale of pain intensity averaged over a week at rest, with a swallow, and with a cough. The subjects rated their pain from 0-10 on the pain intensity scale. Scores are reported as means of the pain score with standard deviation.
  This outcome is reported scores collected at the post-surgery visit; 9 to 29 days after the start of study treatment.
Time Frame: Up to 29 days from the start of study treatment
Population: One participant on the Celecoxib Arm withdrew consent from the study treatment before the Post-Operation visit and was not evaluable for this endpoint.
Measure: Mean (Standard Deviation); unit: score on the pain intensity scale
Arm/Group | Celecoxib Arm | Placebo Arm
Number analyzed (Participants) | 4 | 7
score on the pain intensity scale
  While at Rest | 4.63 (2.29) | 1.21 (1.22)
  With a Swallow | 5.00 (2.80) | 1.64 (2.46)
  With a Cough | 4.25 (1.44) | 1.79 (2.80)

3. Secondary Outcome: Assessment of Overall Pain Control and Management for Patients on Celecoxib Compared to Placebo - Pain Control Questionnaire.
Description: Patient satisfaction was assessed with a pain control questionnaire. The participants were asked questions about their pain satisfaction over the last seven days. The pain control questionnaire was scored from 0-100, with smaller values indicating poor pain control satisfaction and larger values indicating excellent pain control satisfaction.
  This outcome was assessed at post-surgery and end of treatment for up to 5 months
Time Frame: post-surgery (up to 29 days from surgery) and end of treatment (up to 5 months from surgery)
Population: One participant on the Celcoxib Arm was not evaluable for this endpoint.
Measure: Mean (Standard Deviation); unit: score on the pain control questionnaire
Arm/Group | Celecoxib Arm | Placebo Arm
Number analyzed (Participants) | 4 | 7
score on the pain control questionnaire
  Post-Operation | 79.86 (17.77) | 96.82 (5.42)
  End of Treatment | 80.55 (21.52) | 88.89 (13.61)

4. Secondary Outcome: Assessment of Overall Pain Control and Management for Patients on Celecoxib Compared to Placebo.
Description: Narcotic consumption was assessed in daily total morphine equivalents averaged over a week. This outcome was assessed at 7 days after surgery and 35 days after surgery.
  Morphine equivalent dose (MED) is the amount of opioid prescription drugs a patient is taking per day. MED is the sum of the total morphine milligram equivalents (MMEs), a common unit for assessing milligrams of morphine, dose per day.
  The Post-Surgery (1-7 days) time point is MED from 1 to 7 days after surgery. The Post-Surgery (1-14 days) time point is MED from 1 to 14 days after surgery. The Post-Surgery (1-26 days) time point is MED from 1 to 26 days after surgery. The Post-Surgery (1-35 days) time point is MED from 1 to 35 days after surgery. The End of Treatment time point is MED from 1 to 146 days after surgery.
Time Frame: Post-Surgery (1-7 days) up to 7 days, Post-Surgery (1-14 days) up to 14 days, Post-Surgery (1-26 days) up to 26 days, Post-Surgery (1-35 days) up to 35 days, and End of Treatment up to 146 days.
Population: One participant on the Celecoxib Arm was not evaluable for this endpoint.
Measure: Mean (Standard Deviation); unit: MME/day
Arm/Group | Celecoxib Arm | Placebo Arm
Number analyzed (Participants) | 4 | 7
MME/day
  Post-Surgery (1-7 days) | 22.19 (22.20) | 28.73 (34.51)
  Post-Surgery (1-14 days) | 14.24 (18.74) | 20.18 (28.78)
  Post-Surgery (1-21 days) | 12.82 (17.21) | 15.85 (25.01)
  Post-Surgery (1-26 days) | 9.88 (15.67) | 13.46 (22.54)
  Post-Surgery (1-35 days) | 8.76 (14.32) | 12.14 (20.91)
  End of Treatment | 6.64 (7.32) | 11.02 (16.96)

5. Secondary Outcome: Assessment of Functional Outcomes for Patients on Celecoxib Compared to Placebo
Description: Assessment of current activity level was assessed utilizing Karnofsky Performance Status (KPS) at the following time points: pre-operation, day 14 of adjuvant therapy, and end of treatment (or last assessment). The KPS is a scale used to measure a subject's ability to perform daily tasks from 100 Normal no complaints no evidence of disease, 50 Requires considerable assistance and frequent medical care, and 0 Dead.
  This assessment was measured at Post-Operation (up to 29 days after surgery), Mid Radiation (up to 112 days after surgery), and End of Treatment (up to 146 days after surgery).
Time Frame: Post-Operation (up to 29 days after surgery), Mid Radiation (up to 112 days after surgery), and End of Treatment (up to 146 days after surgery)
Population: One participant in the Celecoxib Arm was not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Celecoxib Arm | Placebo Arm
Number analyzed (Participants) | 4 | 7
Participants
  Post- Operation: Able to carry on normal activity and to work; no special care needed. | 2 | 5
  Post- Operation: Unable to work; able to live at home & care for personal needs; varying amount of assistance needed. | 2 | 2
  Post- Operation: Unable to care for self; requires institutional or hospital care; disease may be progressing | 0 | 0
  Post- Operation: Not Assessed | 0 | 0
  Mid Radiation: Able to carry on normal activity and to work; no special care needed. | 2 | 2
  Mid Radiation: Unable to work; able to live at home & care for personal needs; varying amount of assistance needed. | 0 | 2
  Mid Radiation: Unable to care for self; requires institutional or hospital care; disease may be progressing | 0 | 0
  Mid Radiation: Not Assessed | 2 | 3
  End of Treatment: Able to carry on normal activity and to work; no special care needed. | 2 | 6
  End of Treatment: Unable to work; able to live at home & care for personal needs; varying amount of assistance needed. | 2 | 1
  End of Treatment: Unable to care for self; requires institutional or hospital care; disease may be progressing | 0 | 0
  End of Treatment: Not Assessed | 0 | 0

6. Secondary Outcome: Assessment of Functional Outcomes for Patients on Celecoxib Compared to Placebo
Description: Assessment of current activity level was assessed utilizing Functional Oral Intake Scale (FOIS) at the following time points: pre-operation, day 14 of adjuvant therapy, and end of treatment (or last assessment).
  FOIS is a standardized scale assessed by the treating investigator to assess the functional level of oral intake in patients with dysphagia. The FOIS measures from 1 (Aspirates saliva, Nothing by mouth),2 (Tube dependent, Nothing by mouth/minimal trials), 3 (Tube dependent, Full trials by mouth), 4 (Total Oral Single, texture trials), 5 (Total Oral, Multiple texture trials), 6 (Total Oral, By mouth/ restrictions Minimal), and 7 (Regular diet, By mouth/ no restrictions). This assessment was measured for up to 5 months.
  This assessment was measured at Post-Operation (up to 29 days after surgery), Mid Radiation (up to 112 days after surgery), and End of Treatment (up to 146 days after surgery).
Time Frame: as for outcome 5
Population: One participant on the Celecoxib Arm was not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Celecoxib Arm | Placebo Arm
Number analyzed (Participants) | 4 | 7
Participants
  Post-Operation: Aspirates Saliva | 0 | 0
  Post-Operation: Tube Dependent | 1 | 2
  Post-Operation: Total Oral | 3 | 4
  Post-Operation: Regular Diet | 0 | 1
  Post-Operation: Not Assessed | 0 | 0
  Mid-Radiation: Aspirates Saliva | 0 | 0
  Mid-Radiation: Tube Dependent | 1 | 2
  Mid-Radiation: Total Oral | 1 | 2
  Mid-Radiation: Regular Diet | 0 | 0
  Mid-Radiation: Not Assessed | 2 | 3
  End of Treatment (or last assessment): Aspirates Saliva | 0 | 0
  End of Treatment (or last assessment): Tube Dependent | 1 | 1
  End of Treatment (or last assessment): Total Oral | 3 | 2
  End of Treatment (or last assessment): Regular Diet | 0 | 4
  End of Treatment (or last assessment): Not Assessed | 0 | 0

7. Secondary Outcome: Assessment of Functional Outcomes for Patients on Celecoxib Compared to Placebo
Description: Assessment of swallowing capabilities was assessed by determining gastrostomy tube (G-tube) utilization at the following time points: pre-operation, day 14 of adjuvant therapy, and end of treatment (or last assessment). A G-tube is a tube inserted surgically through the abdomen and into the stomach to deliver liquids, medications, and nutrients directly into the stomach.
  The responses in this outcome measure are Yes (G-tube is being utilized), No (G-tube is not being utilized), and Not Assessed (G-tube utilized was not assessed).
  This assessment was measured at Post-Operation (up to 29 days after surgery), Mid Radiation (up to 112 days after surgery), and End of Treatment (up to 146 days after surgery).
Time Frame: as for outcome 5
Population: One participant on the Celecoxib Arm was not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Celecoxib Arm | Placebo Arm
Number analyzed (Participants) | 4 | 7
Participants
  Post-Operation: Yes | 1 | 2
  Post-Operation: No | 3 | 5
  Post-Operation: Not Assessed | 0 | 0
  Mid-Radiation: Yes | 1 | 2
  Mid-Radiation: No | 1 | 2
  Mid-Radiation: Not Assessed | 2 | 3
  End of Treatment (or Last Assessment): Yes | 2 | 1
  End of Treatment (or Last Assessment): No | 2 | 6
  End of Treatment (or Last Assessment): Not Assessed | 0 | 0

8. Secondary Outcome: To Assess the Effect of Celecoxib Therapy on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Head and Neck Module (EORTC QLQ-HN43) Compared to Placebo.
Description: The EORTC QLQ-HN43 is a 43-question assessment for determining the health-related quality of life of head and neck cancer patients participating in clinical trials. Patients indicate which symptoms/problems they have experienced during the past week, from "1 Not at All" to "4 Very Much".
  The assessment was scored according to the "EORTC QLQ-C30 Scoring Manual", reporting data as 19 subscales with scores from 0-100. A high scale score represents a higher response level.
  A high functional scale score (FS) represent a high/healthy level of function and includes body image, social contact, & sexuality A high symptom scale score (SS) represent a high level of symptomatology/problems and includes anxiety, cough, head and neck pain, swallowing, neurologic problems, senses, speech, social eating, weight loss, problems w/ skin, shoulder, wound healing, dry mouth, opening mouth, neck swelling, & teeth.
  This outcome will report the mean score of each subscale.
Time Frame: Up to 29 days after surgery (up to 32 days after initiation of study treatment)
Population: One participant on Arm 1 withdrew consent from the study treatment before the Post-Operation visit and was not evaluable for this endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Celecoxib Arm | Placebo Arm
Number analyzed (Participants) | 4 | 7
units on a scale
  Anxiety (SS) | 50 (36) | 50 (34.69)
  Body Image (FS) | 36.11 (31.91) | 60.32 (34.46)
  Coughing (SS) | 16.67 (19.25) | 9.52 (16.27)
  Dry mouth and sticky saliva (SS) | 54.17 (31.55) | 42.86 (33.13)
  Neurological problems (SS) | 44.44 (50.92) | 9.52 (16.27)
  Opening mouth (SS) | 66.67 (47.14) | 42.86 (25.20)
  Pain in the head and neck (SS) | 41.67 (20.41) | 27.38 (28.35)
  Social contact (FS) | 50 (19.25) | 61.90 (35.63)
  Problems with senses (SS) | 25 (21.52) | 28.57 (35.63)
  Shoulder problems (SS) | 45.83 (45.90) | 9.52 (13.11)
  Skin problems (SS) | 25 (13.98) | 20.63 (31.71)
  Swelling in the neck (SS) | 66.67 (47.14) | 57.14 (46)
  Social eating (SS) | 50 (43.3) | 26.19 (29.83)
  Speech problems (SS) | 55.24 (26.15) | 48.10 (34.53)
  Problems with Swallowing (SS) | 45.83 (29.46) | 29.76 (33.97)
  Problems with Sexuality (FS) | 33.33 (33.33) | 80.95 (26.23)
  Problems with teeth (SS) | 22.22 (27.22) | 22.22 (24.84)
  Weight loss (SS) | 25 (16.67) | 14.29 (26.23)
  Problems with wound healing (SS) | 33.33 (47.14) | 28.57 (23)

9. Secondary Outcome: To Assess the Effect of Celecoxib Therapy on the MDASI-HN Questionnaire Compared to Placebo.
Description: This outcome will report the quality of life questionnaire, the M. D. Anderson symptom inventory head neck (MDASI-HN) at the Post-Operation Visit. This was assessed up to 29 days after surgery (up to 32 days after initiation of study treatment).
  MDASI-HN is a 28-question, 2-part questionnaire for patients with head and neck cancer that assesses the severity of symptoms and impact on daily life. In Part I, subjects indicated how severe their symptoms were from "0 Not present" to "10 As Bad as You can Imagine". In Part II, subjects indicated how symptoms have interfered with their live from "0 Did not Interfere" to "10 Interfered Completely".
  This assessment was scored according to the The M. D. Anderson Symptom Inventory User Guide.
Time Frame: Up to 29 days after surgery (up to 32 days after initiation of study treatment)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Celecoxib Arm | Placebo Arm
Number analyzed (Participants) | 4 | 7
points
  General Symptom Factor | 4.48 (2.00) | 3.06 (2.12)
  Gastrointestinal Symptoms Factor | 1.92 (1.29) | 1.76 (2.45)
  HNC Symptoms | 6.23 (2.60) | 3.39 (2.62)
  HNC Treatment-Related Symptoms | 3.55 (1.81) | 1.60 (2.05)
  General Cancer Related Symptoms | 3.88 (1.70) | 2.75 (2.12)
  Head and Neck Cancer Related Symptoms | 4.58 (1.92) | 2.37 (1.84)
  Symptoms Interference with Daily Activities | 6.42 (2.18) | 4.45 (2.66)

10. Secondary Outcome: Assessment of the Average Number of Treatment Days Missed During Adjuvant Radiation for Patients on Celecoxib Compared to Placebo.
Description: This outcome will report the number of participants who missed treatment days during adjuvant radiation, who did not miss any treatment days during adjuvant radiation, and the number of participants who did not start adjuvant radiation therapy.
Time Frame: up to 140 days
Population: One participant on the Celecoxib Arm was not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Celecoxib Arm | Placebo Arm
Number analyzed (Participants) | 4 | 7
Participants
  No Adjuvant Radiation Therapy | 2 | 1
  No days of missed adjuvant radiation therapy | 2 | 5
  More than 0 days of adjuvant radiation therapy | 0 | 1

ADVERSE EVENTS:
Time Frame: Collection of adverse events began on the first dose of study medication until the end of treatment visit (or until a new cancer treatment is initiated). Adverse events were collected for up to 5 months.
Arm/Group | Celecoxib Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/7
Serious Adverse Events (participants affected / at risk) | 2/5 | 1/7
Other Adverse Events (participants affected / at risk) | 5/5 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Celecoxib Arm (N=5) | Placebo Arm (N=7)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Celecoxib Arm (N=5) | Placebo Arm (N=7)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (5) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (3) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2) | 1 (1)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (4) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (3) | 2 (3)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 2 (4) | 2 (2)
Pain (General disorders) | 2 (3) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) | 1 (2)
Thrush (Infections and infestations) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0)
Weight loss (Investigations) | 1 (2) | 2 (3)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-18): https://cdn.clinicaltrials.gov/large-docs/73/NCT04162873/Prot_SAP_000.pdf